CLINICAL TRIAL: NCT04721977
Title: A Phase 2 Open-label, Single Arm Study of MK-7119 in Combination With Trastuzumab and Capecitabine in Participants With Previously Treated Locally Advanced Unresectable or Metastatic HER2+ Breast Carcinoma
Brief Title: A Study of Tucatinib (MK-7119) in Combination With Trastuzumab and Capecitabine in Participants With Previously Treated Locally Advanced Unresectable or Metastatic Human Epidermal Growth Factor Receptor 2 Positive (HER2+) Breast Carcinoma (MK-7119-001)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7119-001; MK-7119-001 (Other: Merck); jRCT2051200152 (Registry Identifier: jRCT)
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — tucatinib; Trastuzumab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tucatinib + Trastuzumab + Capecitabine (Experimental): Participants will receive tucatinib plus trastuzumab plus capecitabine. Tucatinib 300 mg will be administered orally twice daily (BID). Trastuzumab 8 mg/kg loading dose followed by 6 mg/kg maintenance dose thereafter, will be administered intravenously (IV) on Day 1 of each 21-day cycle. Capecitabine 1000 mg/m^2 will be administered orally BID on Days 1-14 of each 21-day cycle. Tucatinib, trastuzumab and capecitabine treatment will continue until unacceptable toxicity, disease progression, death, withdrawal of consent or study closure.
  Interventions: Drug: Tucatinib; Biological: Trastuzumab; Drug: Capecitabine

INTERVENTIONS:
Drug: Tucatinib — Tucatinib 300 mg administered BID via oral tablet
  Other Names: MK-7119; Tukysa
Biological: Trastuzumab — Trastuzumab 8 mg/kg loading dose followed by 6 mg/kg maintenance dose, administered via IV infusion
  Other Names: Herceptin; Herceptin Hylecta
Drug: Capecitabine — Capecitabine 1000 mg/m^2 administered BID via oral tablet
  Other Names: Xeloda

SUMMARY:
The goal of this study is to evaluate the efficacy and safety of tucatinib in combination with trastuzumab and capecitabine in participants with unresectable locally advanced or metastatic HER2+ breast cancer who have had prior treatment with taxane anti-cancer agent, trastuzumab, pertuzumab and trastuzumab emtansine (T-DM1). The primary hypothesis is that the confirmed objective response rate (cORR) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) as determined by independent central review (ICR) for the combination of tucatinib, trastuzumab and capecitabine, is greater than 20%.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically confirmed HER2+ breast carcinoma
* Has received previous treatment with taxane anti-cancer agent, trastuzumab, pertuzumab, and T-DM1 with the exception of when the use of taxanes is contraindicated or judged not to be the best treatment at the investigator's discretion
* Has radiographically and/or histologically confirmed disease progression on last systemic anticancer treatment
* Has adequate organ function
* Female participant is not pregnant or breastfeeding and is not a woman of childbearing potential (WOCBP) or is a WOCBP and using contraception or abstinent from heterosexual intercourse during the intervention period and for at least 30 days after receiving the last dose of tucatinib, 80 days after receiving the last dose of trastuzumab, or 180 days after receiving the last dose of capecitabine, whichever occurs last and agrees to not donate eggs during this period
* Male participants refrain from donating sperm and are either abstinent from heterosexual intercourse or agree to use contraception during the intervention period and for at least 7 days after receiving the last dose of tucatinib and 90 days after receiving the last dose of capecitabine, whichever occurs last
* Previously treated brain metastasis is stable or progressed, provided there is no clinical indication for immediate re-treatment

Exclusion Criteria:

* Has been previously treated with lapatinib within 12 months of starting study treatment
* Has been previously treated with neratinib, afatinib, tucatinib or capecitabine
* Has a history of exposure to doxorubicin, epirubicin, mitoxantrone, idarubicin, liposomal doxorubicin
* Has had treatment with any systemic anti-cancer therapy including hormonal therapy, non-central nervous system (CNS) radiation or experimental agent ≤3 weeks before first dose of study treatment
* Has any toxicity related to prior cancer therapies that has not resolved with the exception of alopecia, congestive heart failure, anemia
* Has clinically significant cardiopulmonary disease
* Has known myocardial infarction or unstable angina within 6 months prior to the first dose of study treatment
* Has any uncontrolled viral, bacterial or fungal infection within 14 days prior to the first dose of study treatment
* Is positive for Hepatitis B, Hepatitis C or has known chronic liver disease
* Is known to be positive for human immunodeficiency virus (HIV)
* Has evidence within 2 years of the start of study treatment of another malignancy that required systemic treatment
* Has ongoing use of systemic corticosteroids for control of symptoms of brain metastases
* Has any brain lesion thought to require immediate local therapy
* Has known or suspected leptomeningeal disease (LMD)
* Has poorly controlled generalized or complex partial seizures or manifest neurologic progression due to brain metastases

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2026-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (28):
- Japan (24):
  - Aichi Cancer Center Hospital ( Site 1013), Nagoya, Aichi-ken
  - Nagoya University Hospital ( Site 1021), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 1002), Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center ( Site 1014), Matsuyama, Ehime
  - National Hospital Organization Hokkaido Cancer Center ( Site 1017), Sapporo, Hokkaido
  - Hokkaido University Hospital ( Site 1022), Sapporo, Hokkaido
  - Hyogo Cancer Center ( Site 1005), Akashi, Hyōgo
  - Hyogo College of Medicine Hospital ( Site 1019), Nishinomiya, Hyōgo
  - University of Tsukuba Hospital ( Site 1020), Tsukuba, Ibaraki
  - Kanagawa Cancer Center ( Site 1010), Yokohama, Kanagawa
  - Medical Corporation Nahanishikai Nahanishi Clinic ( Site 1016), Naha, Okinawa
  - Saitama Cancer Center ( Site 1018), Kitaadachi-gun, Saitama
  - National Hospital Organization Kyushu Cancer Center ( Site 1009), Fukuoka
  - Fukushima Medical University Hospital ( Site 1012), Fukushima
  - Hiroshima City Hiroshima Citizens Hospital ( Site 1024), Hiroshima
  - Social medical corporation Hakuaikai Sagara Hospital ( Site 1008), Kagoshima
  - Kumamoto Shinto General Hospital ( Site 1007), Kumamoto
  - National Hospital Organization Osaka National Hospital ( Site 1001), Osaka
  - Osaka International Cancer Institute ( Site 1004), Osaka
  - National Cancer Center Hospital ( Site 1003), Tokyo
  - Juntendo University Hospital ( Site 1025), Tokyo
  - The Cancer Institute Hospital of JFCR ( Site 1015), Tokyo
  - Showa University Hospital ( Site 1023), Tokyo
  - Tokyo Medical University Hospital ( Site 1006), Tokyo
- South Korea (3):
  - Seoul National University Hospital ( Site 2003), Seoul
  - Severance Hospital ( Site 2001), Seoul
  - Samsung Medical Center ( Site 2002), Seoul
- National Cheng Kung University Hospital ( Site 3000), Dawan, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 66 participants were enrolled in this study across Japan, Taiwan and South Korea. Results reported are based on the primary completion date of the study.
Groups:
- Tucatinib + Capecitabine + Trastuzumab: Participants with locally advanced unresectable or metastatic HER2+ breast cancer who have had prior treatment with taxane anti-cancer agent, trastuzumab, pertuzumab, and trastuzumab emtansine (T-DM1) were administered Tucatinib 300 mg tablets orally BID, Capecitabine tablets 1000 mg/m^2 orally BID on Days 1 to 14 of each 21-day cycle and Trastuzumab was administered as a loading dose of 8 mg/kg IV followed by 6 mg/kg once every 21 days until unacceptable toxicity, disease progression, death, withdrawal of consent, or study closure.
Period: Overall Study
Arm/Group | Tucatinib + Capecitabine + Trastuzumab
Started | 66
Japanese Participants | 53
Completed | 0
Not Completed | 66
Not completed — Death | 15
Not completed — Ongoing | 51

BASELINE CHARACTERISTICS:
Population: All treated participants set included all participants who received any amount of study drug.
Arm/Group | Tucatinib + Capecitabine + Trastuzumab
Number analyzed (Participants) | 66
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.6 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 66
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic, Latino/a, or of Spanish Origin | 66

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Objective Response Rate(cORR) Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 Determined by Independent Central Review (ICR): Japanese Participants
Description: cORR was defined as percentage of participants with confirmed complete response (CR) or partial response (PR), per RECIST version 1.1. CR: disappearance of all target lesions. Any pathological lymph nodes must have a reduction in short axis to <10 millimeter(mm). PR: a >=30% decrease in the sum of diameters of target lesions, taking as a reference the baseline sum diameters. Only response assessments before first documented progressive disease(PD) or new anti-cancer therapies were considered. PD: at least a 20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study(included baseline sum if smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Appearance of one or more new lesions was also considered PD. Participants with missing data were considered non-responders. cORR was determined by ICR. Two-sided 90% exact confidence interval was based on Clopper-Pearson method.
Time Frame: From date of first dose until first documented disease progression or start of new anticancer therapy, whichever occurred first (maximum up to 17.8 months)
Population: Response evaluable set for Japanese population included all Japanese participants enrolled in Japanese sites who met all of the following criteria: (1) had measurable disease at baseline, (2) received any amount of study treatment, and (3) had at least one post baseline disease assessment or discontinued due to clinical progression, toxicity, or death. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Tucatinib + Capecitabine + Trastuzumab
Number analyzed (Participants) | 48
Percentage of participants | 35.4 [24.0 to 48.3]

2. Secondary Outcome: Confirmed Objective Response Rate(cORR) Per RECIST Version 1.1 Determined by ICR: All Participants
Description: cORR was defined as percentage of participants with confirmed CR or PR, per RECIST version 1.1. CR: disappearance of all target lesions. Any pathological lymph nodes must have a reduction in short axis to <10 mm. PR: a >=30% decrease in the sum of diameters of target lesions, taking as a reference the baseline sum diameters. Only response assessments before first documented PD or new anti-cancer therapies were considered. PD: at least a 20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study (included baseline sum if smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Appearance of one or more new lesions was also considered PD. Participants with missing data were considered non-responders. cORR was determined by ICR. Two-sided 90% exact confidence interval was based on Clopper-Pearson method.
Time Frame: From date of first dose until first documented disease progression or start of new anticancer therapy, whichever occurred first
Reporting Status: Not Posted, anticipated posting 2028-12

3. Secondary Outcome: Confirmed Objective Response Rate(cORR) Per RECIST Version 1.1 Determined by Investigator Assessment (INV): Japanese Participants
Description: cORR was defined as percentage of participants with confirmed CR or PR, per RECIST version 1.1. CR: disappearance of all target lesions. Any pathological lymph nodes must have a reduction in short axis to <10 mm. PR: a >=30% decrease in the sum of diameters of target lesions, taking as a reference the baseline sum diameters. Only response assessments before first documented PD or new anti-cancer therapies were considered. PD: at least a 20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study (included baseline sum if smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Appearance of one or more new lesions was also considered PD. Participants with missing data were considered non-responders. cORR was determined by INV. Two-sided 90% exact confidence interval was based on Clopper-Pearson method.
Time Frame: as for outcome 2
Reporting Status: Not Posted, anticipated posting 2028-12

4. Secondary Outcome: Confirmed Objective Response Rate(cORR) Per RECIST Version 1.1 Determined by INV: All Participants
Description: as for outcome 2
Time Frame: as for outcome 2
Reporting Status: Not Posted, anticipated posting 2028-12

5. Secondary Outcome: Duration of Response (DOR) Per RECIST Version 1.1 Determined by INV: All Participants
Description: DOR was defined as the time from the first objective response (CR or PR that is subsequently confirmed) to documented PD per RECIST version 1.1 or death from any cause, whichever occurred first. CR: disappearance of all target lesions. Any pathological lymph nodes must have a reduction in short axis to <10 mm. PR: a >=30% decrease in the sum of diameters of target lesions, taking as a reference the baseline sum diameters. Only response assessments before first documented PD or new anti-cancer therapies were considered. PD: at least a 20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study (included baseline sum if smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Appearance of one or more new lesions was also considered PD. Only those participants who achieved a confirmed response will be included in the analysis. DOR was determined by INV.
Time Frame: From date of first objective response (CR or PR that is subsequently confirmed) to documented PD, or death from any cause whichever occurred first
Reporting Status: Not Posted, anticipated posting 2028-12

6. Secondary Outcome: Duration of Response (DOR) Per RECIST Version 1.1 Determined by INV: Japanese Participants
Description: as for outcome 5
Time Frame: as for outcome 5
Reporting Status: Not Posted, anticipated posting 2028-12

7. Secondary Outcome: Duration of Response (DOR) Per RECIST Version 1.1 Determined by ICR: All Participants
Description: DOR was defined as the time from the first objective response (CR or PR that is subsequently confirmed) to documented PD per RECIST version 1.1 or death from any cause, whichever occurred first. CR: disappearance of all target lesions. Any pathological lymph nodes must have a reduction in short axis to <10 mm. PR: a >=30% decrease in the sum of diameters of target lesions, taking as a reference the baseline sum diameters. Only response assessments before first documented PD or new anti-cancer therapies were considered. PD: at least a 20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study (included baseline sum if smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Appearance of one or more new lesions was also considered PD. Only those participants who achieved a confirmed response will be included in the analysis. DOR was determined by ICR.
Time Frame: as for outcome 5
Reporting Status: Not Posted, anticipated posting 2028-12

8. Secondary Outcome: Duration of Response (DOR) Per RECIST Version 1.1 Determined by ICR: Japanese Participants
Description: as for outcome 7
Time Frame: as for outcome 5
Reporting Status: Not Posted, anticipated posting 2028-12

9. Secondary Outcome: Progression Free Survival (PFS) Per RECIST Version 1.1 Determined by ICR: All Participants
Description: PFS time was defined as the time from the first date of study treatment to the date of documented disease progression using RECIST v1.1 or death from any cause, whichever occurred first. Participants who were alive and had not progressed at the time of the analysis were censored at the time of their last tumor assessment documenting absence of PD. Participants lacking an evaluation of tumor response after their start of study treatment had their event time censored at 1 day. PD: at least a 20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study (included baseline sum if smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Appearance of one or more new lesions was also considered PD. PFS was determined by ICR.
Time Frame: From date of first dose to the date of documented disease progression or death from any cause whichever occurred first or censoring date
Reporting Status: Not Posted, anticipated posting 2028-12

10. Secondary Outcome: Progression Free Survival (PFS) Per RECIST Version 1.1 Determined by ICR: Japanese Participants
Description: as for outcome 9
Time Frame: as for outcome 9
Reporting Status: Not Posted, anticipated posting 2028-12

11. Secondary Outcome: Progression Free Survival (PFS) Per RECIST Version 1.1 Determined by INV: All Participants
Description: PFS time was defined as the time from the first date of study treatment to the date of documented disease progression using RECIST v1.1 or death from any cause, whichever occurred first. Participants who were alive and had not progressed at the time of the analysis were censored at the time of their last tumor assessment documenting absence of PD. Participants lacking an evaluation of tumor response after their start of study treatment had their event time censored at 1 day. PD: at least a 20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study (included baseline sum if smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Appearance of one or more new lesions was also considered PD. PFS was determined by INV.
Time Frame: as for outcome 9
Reporting Status: Not Posted, anticipated posting 2028-12

12. Secondary Outcome: Progression Free Survival (PFS) Per RECIST Version 1.1 Determined by INV: Japanese Participants
Description: as for outcome 11
Time Frame: as for outcome 9
Reporting Status: Not Posted, anticipated posting 2028-12

13. Secondary Outcome: Overall Survival: All Participants
Description: OS was defined as the time from start of study treatment to date of death due to any cause. In the absence of confirmation of death, survival time was censored at the last date the participant was known to be alive. Participants lacking data beyond their start of study treatment had their survival time censored at 1 day.
Time Frame: From start of study treatment to date of death from any cause or censoring date
Reporting Status: Not Posted, anticipated posting 2028-12

14. Secondary Outcome: Overall Survival: Japanese Participants
Description: as for outcome 13
Time Frame: From start of study treatment to date of death from any cause or censoring date
Reporting Status: Not Posted, anticipated posting 2028-12

15. Secondary Outcome: Number of Participants With Adverse Events, Serious Adverse Events and Treatment Related Adverse Events and Serious Adverse Events: All Participants
Description: An adverse event was defined as any untoward medical occurrence in a participant or clinical investigational participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. Serious adverse event was any untoward medical occurrence at any dose that resulted in death; life-threatening (immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); congenital anomaly/birth defect or that was considered as an important medical event. Treatment related adverse events and serious adverse events was judged by investigator.
Time Frame: From date of first dose of study treatment to up to 30 days after last dose of study treatment
Reporting Status: Not Posted, anticipated posting 2028-12

16. Secondary Outcome: Number of Participants With Adverse Events, Serious Adverse Events and Treatment Related Adverse Events and Serious Adverse Events: Japanese Participants
Description: An adverse event was defined as any untoward medical occurrence in a participant or clinical investigational participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. t intervention indicated and Grade 5 indicates death related to AE. Participants who discontinued treatment due to AEs were captured under AEs leading to treatment discontinuation. SAE was any untoward medical occurrence at any dose that resulted in death; life-threatening (immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); congenital anomaly/birth defect or that was considered as an important medical event. Treatment related adverse events and serious adverse events was judged by investigator.
Time Frame: From date of first dose of study treatment to up to 30 days after last dose of study treatment
Reporting Status: Not Posted, anticipated posting 2028-12

17. Secondary Outcome: Number of Participants With Abnormalities in Laboratory Parameters: All Participants
Time Frame: From date of first dose of study treatment to up to 30 days after last dose of study treatment
Reporting Status: Not Posted, anticipated posting 2028-12

18. Secondary Outcome: Number of Participants With Abnormalities in Laboratory Parameters: Japanese Participants
Time Frame: From date of first dose of study treatment to up to 30 days after last dose of study treatment
Reporting Status: Not Posted, anticipated posting 2028-12

19. Secondary Outcome: Number of Participants With Dose Modifications and Treatment Discontinuations: All Participants
Time Frame: From date of first dose of study treatment to up to 30 days after last dose of study treatment
Reporting Status: Not Posted, anticipated posting 2028-12

20. Secondary Outcome: Number of Participants With Dose Modifications and Treatment Discontinuations: Japanese Participants
Time Frame: From date of first dose of study treatment to up to 30 days after last dose of study treatment
Reporting Status: Not Posted, anticipated posting 2028-12

21. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs: All Participants
Time Frame: From date of first dose of study treatment to up to 30 days after last dose of study treatment
Reporting Status: Not Posted, anticipated posting 2028-12

22. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs: Japanese Participants
Time Frame: From date of first dose of study treatment to up to 30 days after last dose of study treatment
Reporting Status: Not Posted, anticipated posting 2028-12

ADVERSE EVENTS:
Time Frame: From date of first dose of study treatment up to 30 days after last dose of study treatment, death date, or data cut-off date, whichever is earlier (up to 24.6 months)
Description: Same event may appear as both non-SAE and SAE, but what is presented are distinct events. An event may be categorized as serious in 1 participant and non-serious in other participant, or a participant may have experienced both SAE and non-SAE.
Arm/Group | Tucatinib + Capecitabine + Trastuzumab
All-Cause Mortality (participants affected / at risk) | 15/66
Serious Adverse Events (participants affected / at risk) | 6/66
Other Adverse Events (participants affected / at risk) | 65/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tucatinib + Capecitabine + Trastuzumab (N=66)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tucatinib + Capecitabine + Trastuzumab (N=66)
Anaemia (Blood and lymphatic system disorders) | 13 (16)
Abdominal pain upper (Gastrointestinal disorders) | 6 (6)
Cheilitis (Gastrointestinal disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 40 (57)
Nausea (Gastrointestinal disorders) | 32 (41)
Stomatitis (Gastrointestinal disorders) | 18 (19)
Vomiting (Gastrointestinal disorders) | 9 (14)
Fatigue (General disorders) | 9 (13)
Malaise (General disorders) | 13 (18)
Oedema peripheral (General disorders) | 4 (4)
Pyrexia (General disorders) | 8 (9)
Hepatic function abnormal (Hepatobiliary disorders) | 6 (9)
COVID-19 (Infections and infestations) | 9 (9)
Nasopharyngitis (Infections and infestations) | 5 (6)
Paronychia (Infections and infestations) | 10 (10)
Accidental overdose (Injury, poisoning and procedural complications) | 6 (7)
Infusion related reaction (Injury, poisoning and procedural complications) | 5 (5)
Alanine aminotransferase increased (Investigations) | 20 (26)
Aspartate aminotransferase increased (Investigations) | 16 (19)
Blood bilirubin increased (Investigations) | 18 (28)
Blood creatinine increased (Investigations) | 9 (22)
Lymphocyte count decreased (Investigations) | 4 (5)
Neutrophil count decreased (Investigations) | 19 (47)
Platelet count decreased (Investigations) | 7 (12)
Weight decreased (Investigations) | 6 (6)
White blood cell count decreased (Investigations) | 16 (40)
Decreased appetite (Metabolism and nutrition disorders) | 11 (14)
Dysgeusia (Nervous system disorders) | 5 (5)
Headache (Nervous system disorders) | 7 (8)
Renal impairment (Renal and urinary disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (8)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (7)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 41 (43)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2024-02-28): https://cdn.clinicaltrials.gov/large-docs/77/NCT04721977/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT04721977/SAP_001.pdf